CLINICAL TRIAL: NCT05581563
Title: Clinical and Functional Outcomes of Tourniquet Use in Primary Total Knee Arthroplasty
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Mongi Slim Hospital (Other)
Responsible Party: Principal Investigator, mohamed hedi ezzine, Principal Investigator, medical doctor, assistant professor, Mongi Slim Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: mongislim2
Record Dates: First submitted 2022-10-01; First posted 2022-10-14 (Actual); Last update posted 2022-10-14 (Actual); Status verified 2022-10

CONDITIONS: Total Knee Arthroplasty
MeSH Terms: interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Intervention Model Description: Longitudinal Study Designs Cohort Study Simple randomisation with a 1:1 allocation ratio outcomes is measured after tourniquet use
Who Masked: Participant, Outcomes Assessor
Masking Description: the use of general anesthesia of all participants the outcomes assessor will not be able to have any information regarding tourniquet use
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- tourniquet use (Active Comparator): knee replacement surgery with the aid of a tourniquet - a tight band placed around the thigh that restricts blood flow to the knee.
  Interventions: Procedure: total knee arthroplasty(TKA)
- without tourniquet use (Sham Comparator): knee replacement surgery without the aid of a tourniquet - a tight band placed around the thigh that restricts blood flow to the knee.
  Interventions: Procedure: total knee arthroplasty(TKA)

INTERVENTIONS:
Procedure: total knee arthroplasty(TKA) — Knee replacement, also called knee arthroplasty or total knee replacement, is a surgical procedure to resurface a knee damaged by arthritis. Metal and plastic parts are used to cap the ends of the bones that form the knee joint, along with the kneecap. This surgery may be considered for someone who has severe arthritis or a severe knee injury.

SUMMARY:
Many surgeons choose to perform total knee arthroplasty (TKA) surgery with the aid of a tourniquet. A tourniquet is a device that fits around the leg and restricts blood flow to the limb. There is a need to understand whether tourniquets are safe, and if they benefit, or harm, patients. The aim of this study was to determine the benefits and harms of tourniquet use in TKA surgery

DETAILED DESCRIPTION:
randomized controlled trials , comparing TKA with a tourniquet versus without a tourniquet. Outcomes included: post-operative pain measure with analogue visual scale function with Oxford Score , Lysholm score and International Knee Documentation Committee Score intraoperative blood loss measurement of quadriceps tonus in pre- and post-operative according to the international rating measurement of quadriceps area circumference duration of surgery, and length of hospital stay

ELIGIBILITY:
Inclusion Criteria:

* Osteoarthritis Kellgren and Lawrence score III or IV
* Written consent
* Total knee arthroplasty

Exclusion Criteria:

* Neurological dysfunction
* Coagulation disorder
* Glucocorticoids, aspirin, heparin, coumadine, warfarin
* History of pulmonary embolism

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-10-10 (Estimated); Primary Completion 2023-10-10 (Estimated); Study Completion 2023-11-10 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS) | Baseline
  Using a ruler, the score is determined by measuring the distance (mm) on the 10-cm line between the "no pain" anchor and the patient's mark, providing a range of scores from 0-100. A higher score indicates greater pain intensity. Based on the distribution of pain VAS scores in post-surgical patients, mild, moderate, or severe, the following cut points on the pain VAS have been recommended: no pain (0-4 mm), mild pain(5-44 mm), moderate pain (45-74 mm), and severe pain (75-100 mm).
Visual Analogue Scale (VAS) | Day 1
  Using a ruler, the score is determined by measuring the distance (mm) on the 10-cm line between the "no pain" anchor and the patient's mark, providing a range of scores from 0-100. A higher score indicates greater pain intensity. Based on the distribution of pain VAS scores in post-surgical patients, mild, moderate, or severe, the following cut points on the pain VAS have been recommended: no pain (0-4 mm), mild pain(5-44 mm), moderate pain (45-74 mm), and severe pain (75-100 mm).
Visual Analogue Scale (VAS) | Day 2
  Using a ruler, the score is determined by measuring the distance (mm) on the 10-cm line between the "no pain" anchor and the patient's mark, providing a range of scores from 0-100. A higher score indicates greater pain intensity. Based on the distribution of pain VAS scores in post-surgical patients, mild, moderate, or severe, the following cut points on the pain VAS have been recommended: no pain (0-4 mm), mild pain(5-44 mm), moderate pain (45-74 mm), and severe pain (75-100 mm).
International Knee Documentation Committee 2000 | Baseline
  International Knee Documentation Committee (IKDC) 2000 subjective score The score is interpreted as a measure of function such that higher scores represent higher levels of function and lower levels of symptoms. A score of 100 is interpreted to mean no limitation with activities of daily living or sports activities and the absence of symptoms.
International Knee Documentation Committee 2000 | Month 3
  International Knee Documentation Committee (IKDC) 2000 subjective score The score is interpreted as a measure of function such that higher scores represent higher levels of function and lower levels of symptoms. A score of 100 is interpreted to mean no limitation with activities of daily living or sports activities and the absence of symptoms.
International Knee Documentation Committee 2000 | Month 6
  International Knee Documentation Committee (IKDC) 2000 subjective score The score is interpreted as a measure of function such that higher scores represent higher levels of function and lower levels of symptoms. A score of 100 is interpreted to mean no limitation with activities of daily living or sports activities and the absence of symptoms.
Oxford Score (OS) | Baseline
  This score is a patient reported outcome measure that consists of 12 questions about an individual's level of function, activities of daily living and how they have been affected by pain over the preceding four weeks.
  the scoring system from 0-4 where four is the best outcome and total scores range from 0 (poorest function) to 48 (maximal function)
Oxford Score (OS) | Month 3
  This score is a patient reported outcome measure that consists of 12 questions about an individual's level of function, activities of daily living and how they have been affected by pain over the preceding four weeks.
  the scoring system from 0-4 where four is the best outcome and total scores range from 0 (poorest function) to 48 (maximal function)
Oxford Score (OS) | Month 6
  This score is a patient reported outcome measure that consists of 12 questions about an individual's level of function, activities of daily living and how they have been affected by pain over the preceding four weeks.
  the scoring system from 0-4 where four is the best outcome and total scores range from 0 (poorest function) to 48 (maximal function)
Lysholm score | Baseline
  The Lysholm Scale currently consists of eight items that measure: pain (25 points), instability (25 points), locking (15 points), swelling (10 points), limp (5 points), stair climbing (10 points), squatting (5 points), and need for support (5 points). Every question response has been assigned an arbitrary score on an increasing scale. The total score is the sum of each response to the eight questions and may range from 0-100. Higher scores indicate a better outcome with fewer symptoms or disabilities
Lysholm score | Month 3
  The Lysholm Scale currently consists of eight items that measure: pain (25 points), instability (25 points), locking (15 points), swelling (10 points), limp (5 points), stair climbing (10 points), squatting (5 points), and need for support (5 points). Every question response has been assigned an arbitrary score on an increasing scale. The total score is the sum of each response to the eight questions and may range from 0-100. Higher scores indicate a better outcome with fewer symptoms or disabilities
Lysholm score | Month 6
  The Lysholm Scale currently consists of eight items that measure: pain (25 points), instability (25 points), locking (15 points), swelling (10 points), limp (5 points), stair climbing (10 points), squatting (5 points), and need for support (5 points). Every question response has been assigned an arbitrary score on an increasing scale. The total score is the sum of each response to the eight questions and may range from 0-100. Higher scores indicate a better outcome with fewer symptoms or disabilities
perioperative blood loss | Hospital admission to discharge (about 3 days)
  intraoperative blood loss estimation in ml added to postoperative drainage
quadriceps area circumference | Baseline
  Measurement of thigh is usually performed 15 cm proximal to the superior pole of the patella. The thigh circumference is measured in cm with a measurement tape and compared to the normal contralateral knee to determine the amount of quadriceps atrophy present
quadriceps area circumference | Month 3
  Measurement of thigh is usually performed 15 cm proximal to the superior pole of the patella. The thigh circumference is measured in cm with a measurement tape and compared to the normal contralateral knee to determine the amount of quadriceps atrophy present
quadriceps area circumference | Month 6
  Measurement of thigh is usually performed 15 cm proximal to the superior pole of the patella. The thigh circumference is measured in cm with a measurement tape and compared to the normal contralateral knee to determine the amount of quadriceps atrophy present